CLINICAL TRIAL: NCT02365194
Title: Modifying Risk in Ventral Hernia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mike K Liang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-14-1025
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Hernia, Ventral; Weight Loss
Keywords: Ventral Hernia; Prehabilitation
MeSH Terms: conditions — Hernia, Ventral; Weight Loss | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Other): physical conditioning and weight loss intervention done pre-operatively
  Interventions: Behavioral: Prehabilitation
- Standard Counseling (Other): initial clinic counseling
  Interventions: Behavioral: Standard counseling

INTERVENTIONS:
Behavioral: Prehabilitation — information included in arm description
  Arms: Prehabilitation
Behavioral: Standard counseling — information included in arm description
  Arms: Standard Counseling

SUMMARY:
A pre-operative physical conditioning and weight loss intervention (prehabilitation) compared to standard counseling prior to ventral hernia repair for obese patients (BMI 30-40 kg/m2) at a safety-net hospital results in a higher proportion of patients being hernia- and complication-free 2 years after surgical consultation.

DETAILED DESCRIPTION:
Background:

Obesity is a risk factor for ventral hernia complications with or without repair, but the management strategy that best balances overall risks and benefits for obese patients with ventral hernias is unknown. The primary aim of this project is to compare the effect of prehabilitation (preoperative physical conditioning and weight loss intervention) versus standard preoperative counseling followed by repair for obese patients (BMI 30-40 kg/m2) with ventral hernias on outcomes.

Methods:

A comprehensive cohort study of obese patients who have ventral hernias will be performed. Within the comprehensive cohort study, patients who are candidates for elective ventral hernia repair will be randomized to a prehabilitation intervention or standard counseling with surgical repair once weight loss goals have been met. All patients will have repair after 6 months even if they have not met their weight loss goals. Patients who are not eligible for the trial or who refuse to participate will be followed in a non-randomized cohort; they will have their hernia repaired based upon current institution standards. (figure 1) The primary outcome of the study will be proportion of patients who are hernia- and complication- free 2 years after surgical consultation. This composite outcome was chosen in order to encompass all clinically important risks and benefits of both operative and non-operative strategies. Based on power calculations(alpha=0.05, beta=0.20), 232 eligible patients are needed assuming a 30% non-enrollment and 50% dropout. Since this is an efficacy trial, analysis will be performed per protocol as well as intention to treat. The primary outcome will be compared using the Cochran-Mantel-Haenszel test. Generalized linear mixed models (GLMMs) will be used to identify independent predictors of a successful outcome defined as hernia- and complication free at 2 years. In addition to a frequentist analysis, a Bayesian analysis will be performed. Posterior point estimates, credible intervals, and probability of increase in proportion of patients without hernias or complications will be calculated.

Conclusion:

Prehabilitation may have no impact on outcomes following ventral hernia repair, cause more complications with acute hernia presentation, or prove superior and decrease recurrences and complications compared to standard of care. This randomized controlled trial will provide baseline information on the efficacy of prehabiliation prior to open ventral hernia repair in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient desires an elective surgical repair
* Diagnosis of a ventral hernia with width on CT scan of 3-20 cm in diameter
* Age 18 years or greater
* Able to give informed consent
* BMI of 30-40 kg/m2
* Surgical candidate based upon surgeon assessment

Exclusion Criteria:

* Patient has a severe comorbid condition likely to limit survival to < 2 years
* Patient has cirrhosis with or without ascites
* Patient has a bowel obstruction, strangulation, peritonitis, or perforation
* Patient has an indication for urgent surgery determined by surgeon such as full-thickness skin breakdown, enterocutaneous fistula, intermittent incarceration, or severe symptoms
* Patient has a local or systemic infection
* Patient is a prisoner
* Patient is pregnant or intends to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are hernia- and complication-free | 2 years after enrollment

SECONDARY OUTCOMES:
Weight loss (number of participants with weight loss of at least 7%) | 6 months after enrollment
  number of participants with weight loss of at least 7%
Receipt of elective or emergency surgery | 6 months after enrollment
  When the patient underwent elective or emergent surgery
surgery-related complications (number of patients who developed infections or other complications related to the surgery) | 2 years after surgery
  number of patients who developed infections or other complications related to the surgery
hernia-related complications (number of patients who developed complications from their hernia) | 2 years after surgery
  number of patients who developed complications from their hernia
Functional Status (Quality of life questionnaire responses) | 2 years after surgery
  Quality of life questionnaire responses
implementation outcomes (difference in costs between the patients in the treatment group and those in the usual care group) | 2 years
  difference in costs between the patients in the treatment group and those in the usual care group
Physiologic changes (number of pounds lost/gained) | 2 years after surgery
  number of pounds lost/gained
Metabolic changes (difference in basal metabolic rate before treatment and after treatment) | 2 years after surgery
  difference in basal metabolic rate before treatment and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mike K Liang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Bernardi K, Olavarria OA, Dhanani NH, Lyons N, Holihan JL, Cherla DV, Berger DH, Ko TC, Kao LS, Liang MK. Two-year Outcomes of Prehabilitation Among Obese Patients With Ventral Hernias: A Randomized Controlled Trial (NCT02365194). Ann Surg. 2022 Feb 1;275(2):288-294. doi: 10.1097/SLA.0000000000004486. PMID 33201119
- [Derived] Liang MK, Bernardi K, Holihan JL, Cherla DV, Escamilla R, Lew DF, Berger DH, Ko TC, Kao LS. Modifying Risks in Ventral Hernia Patients With Prehabilitation: A Randomized Controlled Trial. Ann Surg. 2018 Oct;268(4):674-680. doi: 10.1097/SLA.0000000000002961. PMID 30048306